CLINICAL TRIAL: NCT03587441
Title: The Efficacy of Neostigmine as an Adjuvant to Bupivacaine for Intrathecal Block in Reducing the Incidence and Severity of Post-Dural Puncture Headache for Parturients Scheduled for Elective Caesarean Section
Brief Title: Intrathecal Neostigmine for Prevention of PDPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany M Yassin, MD, Associate Professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M335
Record Dates: First submitted 2018-06-13; First posted 2018-07-16 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Post-Dural Puncture Headache
Keywords: postural headache; intrathecal neostigmine for prevention of PDPH
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Neostigmine; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Intervention Group (N) (Active Comparator): Neostigmine Methylsulfate intervention : A one milliliter syringe will contain 20 µg of Neostigmine methyl sulfate. 0.5 mg ampule (1 ml) will be diluted in 4 ml dextrose 5% to make a solution of 100 µg/ml, 0.2 ml of this solution will be added to 2.5 ml of hyperbaric bupivacaine 0.5 % used for intrathecal injection.
  Interventions: Drug: Neostigmine Methylsulfate; Drug: Dextrose 5% in water
- The Control Group (P) (Placebo Comparator): Dextrose 5% in water intervention : an equal volume (0.2 ml) of dextrose 5% will be added to 2.5 ml of hyperbaric bupivacaine 0.5 % used for intrathecal injection.
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Neostigmine Methylsulfate — 20 µg Neostigmine Methylsulfate intrathecal in 0.2 ml of Dextrose 5% solution
  Other Names: Neostigmine (0.5 mg)
  Arms: The Intervention Group (N)
Drug: Dextrose 5% in water — intrathecal
  Other Names: Dextrose 5% in Water (D5W)

SUMMARY:
Neuraxial blocks continue to be the cornerstone of anesthesia and postoperative analgesia for normal vaginal delivery and elective caesarean section due to its approved safety and efficiency for decades. Post-dural puncture headache (PDPH) is still one of the most common complications of neuraxial anesthetic techniques. The headache could be severe and limit the activities of the new mother to care for her baby, prolong hospital stay.

PDPH is defined as a headache that develops within five days of dural puncture and can't be attributed to any other types of headache and mostly is postural in character.

Neostigmine methylsulfate is a synthetic carbamic acid ester which reversibly inhibits the enzyme Acetylcholine esterase (AChE) that makes more Acetylcholine molecules available at cholinergic receptors. Neostigmine is used in anesthesia mainly as a reversal for non-depolarizing neuromuscular agents.

Intrathecal (IT) neostigmine was tried as an adjuvant to local anesthetics in IT block for elective cesarean sections to decrease local anesthetic consumption and to prolong postoperative analgesia. Side effects of IT neostigmine are dose-dependent with doses more than 25 µg especially nausea and vomiting and could be decreased by increasing the baricities of the local anesthetic solutions and by early head up position after IT injection. However, its effect on PDPH was not investigated before in literature.

Parturients will be randomly assigned into one of two groups: the intervention group will receive 20 µg with IT Bupivacaine and the control group will receive an equivalent volume of dextrose 5% with the IT Bupivacaine.

The objective of the current study is to evaluate the efficacy and safety of IT neostigmine as an adjuvant to bupivacaine in reducing the incidence and severity of post-dural puncture headache in parturients scheduled for an elective cesarean section.

DETAILED DESCRIPTION:
The study will be performed from July 2018 to July 2019 at Fayoum University hospital after approval of the local institutional ethics committee and local institutional review board. The study design will be prospective, randomized, double-blind, parallel groups, placebo-controlled clinical trial. A detailed informed consent will be signed by the eligible participants before recruitment and randomization.

Randomization will be done by using computer-generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before IT block. Neither the participants, the study investigators, the attending clinicians, nor the data collectors will be aware of groups' allocation until the study end. The Consolidated Standards of Reporting Trials (CONSORT) recommendations for reporting randomized, controlled clinical trials will be followed.

Preoperative preparations and Premedication:

The study solutions will be prepared in a one milliliter syringe as following: For the intervention group (N), it will contain 20 µg of Neostigmine® (0.5 mg/ml ampules manufactured by Amriya for pharmaceutical industries in Alexandria, Egypt) neostigmine ampule will be diluted in 4 ml dextrose 5% to make a solution of 100 µg/ml, 0.2 ml of this solution will be used, while in the control group an equal volume (0.2 ml) of dextrose 5% will be prepared. The syringes used will be labeled as A and B per their content. The identical coded syringe will be prepared by trained anesthesia technicians who will not be included in the study.

All parturients will receive 150 mg Ranitidine oral tablet on the night before and on the morning of the operation as a premedication.

Intraoperative technique and management:

Upon arrival to the operating room standard monitors (Pulse oximeter, Noninvasive blood pressure monitoring, and Electrocardiogram) will be applied and continued all over the operation, an eighteen gauge (18G) peripheral intravenous (IV) cannula will be inserted, and 10 ml/kg of Ringer lactate solution warmed to 37°C will be infused over 15 minutes as a preload.

IT block will be performed via a midline approach into the L4-5 interspaces in sitting position with complete aseptic condition using a 25 gauge Quincke spinal needle after giving 3 ml of lidocaine 2% (60 mg) as a subcutaneous infiltration. After confirming free cerebrospinal fluid (CSF) flow through the needle a 2.5 ml of hyperbaric bupivacaine 0.5 % in addition to the content of the prepared study syringe will be slowly injected. Then, the parturient will be immediately placed in the supine position with 15° left tilt, and an oxygen mask will be applied at 2 l/min.

After ensuring sufficient anesthesia level, the surgical procedure will start with continuous hemodynamics monitoring and recording. If the systolic blood pressure (SBP) decreased to 20% below the baseline or less than 90 mmHg, ephedrine 5 mg will be administered intravenously. Also, if heart rate (HR) will be less than 50 beats/min, atropine sulfate 0.5 mg will be administered intravenously. Any intraoperative or postoperative nausea or vomiting will be managed with 10 mg of metoclopramide Upon delivery of the fetus, ten units of oxytocin will be given by IV infusion, and if the uterus is not well contracted, additional increments of 5 units will be added accordingly. One gm of Ceftriaxone will be also given after delivery of the fetus by IV infusion.

Postoperative monitoring, Pain control and follow up:

At the end of surgery, Participant will be transferred to postoperative anesthesia care unit (PACU) with standard monitoring applied. All Participants will receive 75 mg diclofenac sodium intramuscular every 12 hours as a pain management per institution policy, 1,23 4 mg of morphine will be given IV if rescue analgesia is needed postoperatively every 10 minutes with a maximum of 20 mg in 6 hours or 32 mg in 24 hours. The participant will be transferred to obstetrics ward after fulfilling the criteria of modified Aldrete scoring system. 24 Assessment for post-dural puncture headache and other associated symptoms will be done from day 0 to day five postoperatively and if the participant will be discharged home, follow up will be done by a phone call. If there will be a complaint of a headache, the participant will be asked to come back to the hospital for proper assessment and management either on an outpatient or inpatient bases per the headache severity.

The participants who will be diagnosed to have PDPH per the criteria of the International Headache Society (HIS) will be treated by using oral medications Panadol extra™ (paracetamol 1gm + caffeine 130 mg) (Manufactured by: Alexandria company for pharmaceuticals & chemical industries under license: GlaxoSmithKline Consumer Healthcare Ltd. Ireland) at 6-hour interval in addition to hydration and bed rest. Severe Intractable headache (VAS ≥ 40) persistent for more than 48 hours with no response to conservative measures will be managed with an epidural blood patch after participant approval and consent signing.

Statistical analysis and sample size estimation:

Continuous variables will be tested for normal distribution by the Shapiro-Wilk test (P ≤ 0.05). Parametric data will be expressed as mean and standard deviation (SD) and analyzed by using the independent t-test. Data with kurtosis or skewness will be depicted as median and interquartile range and compared for significant difference by implementation of Mann-Whitney U test. Categorical variables will be presented as numbers and frequencies and the chi-square test or Fisher exact test will be used to analyze the significant differences between the two arms. A P value ≤ 0.05 will be considered statistically significant. Data will be analyzed using SPSS (SPSS 16.0, SPSS Inc., Chicago, II, USA).

The sample size calculation based on that a 15 % reduction in the incidence of PDPH between the two arms could be of clinically important relevance. The reported incidence of PDPH with the use of 25 gauge Quincke needle is 25 %. Sample size of 100 participants per group were found sufficient assuming (two tail) α = 0.05, β = 0.2 (80 % power), and 1:1 allocation ratio. We will plan to recruit 120 participants per group to account for data loss or protocol violation. The sample size calculation performed with G*Power software version 3.1.9.2 (Institute of Experimental Psychology, Heinrich Heine University, Dusseldorf, Germany).

ELIGIBILITY:
Inclusion Criteria:

* American society association (ASA) physical status II parturients who will be scheduled for an elective caesarean section by IT anesthesia

Exclusion Criteria:

* significant renal, hepatic, and cardiovascular diseases
* pre-eclampsia
* any contraindication to regional anesthesia such as local infection or bleeding disorders
* allergy to neostigmine
* long-term opioid use
* a history of chronic pain, migraine, cluster headache
* digestive problems with nausea or vomiting
* cognitive or memory disorders
* history of urinary retention; bronchial asthma
* perioperative blood transfusion

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
incidence of post-dural puncture headache | At day 5 from intrathecal block
  any headache that develops within five days of dural puncture and can't be attributed to any other types of headache and mostly is postural in character

SECONDARY OUTCOMES:
Visual analog score of post-dural puncture headache (PDPH) at presentation | At 24 hours after headache onset
  Severity of PDPH at presentation estimated by visual analog score (VAS) (where 0 = no headache, and 100 = worst imaginable headache)
Visual analog score of post-dural puncture headache (PDPH) after medical treatment | At 48 hours after starting medical treatment
  Severity of PDPH after 48 hours from receiving medical treatment estimated by visual analog score (VAS) (where 0 = no headache, and 100 = worst imaginable headache)
highest Visual analog score of post-dural puncture headache | At 48 hours after starting medical treatment
  Severity of PDPH estimated by visual analog score (VAS) (where 0 = no headache, and 100 = worst imaginable headache)
Percent of participants with neck stiffness | At 48 hours after headache onset
  incidence of neck stiffness in participants with PDPH in each group
Percent of participants in need for epidural blood patch | After 48 hours from onset of headache
  Severe Intractable headache (VAS ≥ 40) persistent for more than 48 hours with no response to conservative measures will be managed with an epidural blood patch after participant approval and consent signing
Percent of participants complained from intraoperative nausea and vomiting | From intrathecal block until discharge from PACU, assessed up to 24 hours
  Any intraoperative nausea or vomiting related to intrathecal neostigmine injection
Percent of participants complained from postoperative nausea and vomiting | AT 48 hours after PDPH
  Any postoperative nausea or vomiting related to PDPH
incidence of urine retention | At 48 hours from intrathecal block
  postoperative inability to pass urine
incidence of memory and cognitive disorders | At 48 hours from intrathecal block
  any observed or complained memory or cognitive disorders
incidence of hypotension | From intrathecal block until discharge from PACU, assessed up to 24 hours
  systolic blood pressure (≤ 20 % of baseline level or < 90 mmhg
ephedrine requirements | From intrathecal block until discharge from PACU, assessed up to 24 hours
  ephedrine used measured in milligrams
incidence of desaturation | From intrathecal block until discharge from PACU, assessed up to 24 hours
  (SPO2 < 92 %)
incidence of respiratory depression | From intrathecal block until discharge from PACU, assessed up to 24 hours
  Respiratory rate (RR) < 8 bpm
incidence of bradycardia | From intrathecal block until discharge from PACU, assessed up to 24 hours
  heart rate < 50 beat per minute
atropine requirements | From intrathecal block until discharge from PACU, assessed up to 24 hours
  atropine used measured in milligrams
incidence of shivering | From intrathecal block until discharge from PACU, assessed up to 24 hours
  any shivering
time to the first requirement of analgesic supplement | From intrathecal block until discharge from PACU, assessed up to 24 hours
  calculated in minutes
total analgesic consumption | At 24 hour after intrathecal block
  amount of morphine used in milligrams
the assessment of duration of sensory blockade | From intrathecal block until the first appearance of pain at the T10 dermatome, assessed up to 24 hours
  measured in minutes, assessed by a pinprick test
the assessment of duration of motor blockade | From intrathecal block until the modified Bromage score will be zero, assessed up to 24 hours
  measured in minutes, assessed by the modified Bromage score (0, no motor loss; 1, inability to flex the hip; 2, inability to flex the knee; and 3, inability to flex the ankle)
Age | 6 hours before intervention
  in years
Weight | 6 hours before intervention
  in kilograms (kg)
Height | 6 hours before intervention
  in meters (m)
Body mass index | 6 hours before intervention
  in kg/m square
Headache onset | After intrathecal block for five days till appearance of PDPH
  in hours
Duration of surgical procedures | After completion of surgical procedures, within about two hours of intervention
  in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Yassin, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Arevalo-Rodriguez I, Munoz L, Godoy-Casasbuenas N, Ciapponi A, Arevalo JJ, Boogaard S, Roque I Figuls M. Needle gauge and tip designs for preventing post-dural puncture headache (PDPH). Cochrane Database Syst Rev. 2017 Apr 7;4(4):CD010807. doi: 10.1002/14651858.CD010807.pub2. PMID 28388808
- [Background] Nath S, Koziarz A, Badhiwala JH, Alhazzani W, Jaeschke R, Sharma S, Banfield L, Shoamanesh A, Singh S, Nassiri F, Oczkowski W, Belley-Cote E, Truant R, Reddy K, Meade MO, Farrokhyar F, Bala MM, Alshamsi F, Krag M, Etxeandia-Ikobaltzeta I, Kunz R, Nishida O, Matouk C, Selim M, Rhodes A, Hawryluk G, Almenawer SA. Atraumatic versus conventional lumbar puncture needles: a systematic review and meta-analysis. Lancet. 2018 Mar 24;391(10126):1197-1204. doi: 10.1016/S0140-6736(17)32451-0. Epub 2017 Dec 7. PMID 29223694
- [Background] Fattahi Z, Hadavi SM, Sahmeddini MA. Effect of ondansetron on post-dural puncture headache (PDPH) in parturients undergoing cesarean section: a double-blind randomized placebo-controlled study. J Anesth. 2015 Oct;29(5):702-7. doi: 10.1007/s00540-015-2000-5. Epub 2015 Mar 27. PMID 25812804
- [Background] Cossu AP, De Giudici LM, Piras D, Mura P, Scanu M, Cossu M, Saba M, Finco G, Brazzi L. A systematic review of the effects of adding neostigmine to local anesthetics for neuraxial administration in obstetric anesthesia and analgesia. Int J Obstet Anesth. 2015 Aug;24(3):237-46. doi: 10.1016/j.ijoa.2015.05.002. Epub 2015 May 19. PMID 26119258